CLINICAL TRIAL: NCT04933045
Title: Treatment of Syndesmotic Disruption With Anatomic Distal Tibiofibular Ligament Augmentation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. Clair Orthopaedics (Other)
Responsible Party: Principal Investigator, Christopher N Zingas, Orthopedic Surgeon, St. Clair Orthopaedics
Other Study IDs: Syndesmotic Augmentation
Record Dates: First submitted 2021-06-13; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Syndesmotic Injuries
Keywords: Syndesmosis
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Syndesmotic Fixation Group: Cohort of patients treated with anatomic ATFL reconstruction for syndesmotic ankle injury.
  Interventions: Device: Arthrex InternalBrace

INTERVENTIONS:
Device: Arthrex InternalBrace — Placement of Arthrex InternalBrace for anatomic distal tibiofibular ligament augmentation to stabilize the ankle syndesmosis during surgery.

SUMMARY:
The primary objective is to evaluate indications and outcomes of operative fixation of syndesmotic injuries, at least in part, with direct anatomic augmentation in acute and subacute traumatic cases. The secondary objective of the study is to evaluate clinically the InternalBraceTm to facilitate the direct syndesmotic fixation/augmentation.

DETAILED DESCRIPTION:
A syndesmosis is a slightly movable fibrous joint in which bones such as the tibia and fibula are joined together by connnective tissue. Together, they form a bracket shaped socket, covered in hyaline cartilage. This socket is known as the mortise. A syndesmotic or 'high 'ankle sprain is when the ligaments binding the distal tibia and fibula at the ankle joint are injured or torn. This can lead to the ankle joint and syndesmoses to being malaligned, subluxed or widened. Subsequently, this can lead to ankle arthritis and deformity with persistent pain and swelling about the ankle.

There are no generally accepted treatment guidelines. Thus, there still remains considerable controversies regarding diagnosis, classification and treatment of syndesmotic injuries. Syndesmotic malreduction is the most common indication for early re-operation after ankle fracture surgery, and widening of the ankle mortise by only 1 mm decreases the contact area of the tibiotalar joint by 42%. Outcome of ankle fractures with syndesmosis injury is worse than without, even after surgical syndesmotic stabilization. This may be due to a high incidence of syndesmotic malreduction revealed by increasing postoperative computed tomography controls. Therefore, even open visualization of the syndesmosis during the reduction maneuver has been recommended. Thus, the most important clinical predictor of outcome is consistently reported as accuracy of anatomic reduction of the injured syndesmosis. In 2017 a new syndesmotic InternalBraceTM technique for improved anatomic distal tibiofibular ligament augmentation to protect healing of the injured native ligaments was introduced. This technique involves direct surgical inspection of the syndesmoses for injury and subsequent augmentation.

This study hopes to evaluate the results of this direct syndesmotic augmentation/stabilization to help determine if this is perhaps a safer, and possibly more effective method.

This prospective study is designed to evaluate 32 consecutive patients that did have an acute or subacute syndesmotic injury that necessitated surgical stabilization and used at least in part the InternalBrace technique. There was not a restriction of age, gender, or race.

2 patients who were labeled as having severe syndesmotic disruption and had additional screw fixation. Also, 5 patients had dynamic syndesmotic fixation in addition to direct InternalBrace augmentation of the AITFL.

The patents will or had had plain radiographs and physical examination of injured ankle 1 week, 1 month, 3 months, 6 months and 12 months. Also, at minimum 12 months post operatively a physical exam and plain radiograph contralateral uninjured ankle to be performed as comparison/control. At minimum 12 months post operative additional patent report outcomes such as AOFAS/VAS scores and return to pre-injury status recreationally/work level to be evaluated. The ankle anatomic syndesomotic and mortise alignment has been associated with long term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients that occurred an ankle syndesmotic injury necessitating surgical stabilization/fixation

Exclusion Criteria:

* Skeletally immature patients, patients with nonoperatively managed ankle injuries

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Skeletally mature patients that occurred an ankle syndesmotic injury necessitating surgical stabilization/fixation
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Indications and outcomes of operative fixation of syndesmotic injuries | 1 year
  Evaluate indicatinos and outcomes of operative fixation of syndesmotic injuries at least in part with direct anatomic augmentation in acute and subacute traumatic ankle fracture cases.

SECONDARY OUTCOMES:
InternalBrace | 1 yeaer
  Evaluate clinically the InternalBrace to facilitate the direct syndesmotic fixation/augmentation.

CONTACTS AND LOCATIONS:
Locations (1):
- St Clair Orthopedics and Sports Medicine, Saint Clair Shores, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided